CLINICAL TRIAL: NCT01891383
Title: Endophenotypes of Dementia Associated With Traumatic Brain Injury in Retired Military Personnel
Brief Title: Clinical Characteristics of Dementias That Occur Remotely After Traumatic Brain Injury in Retired Military Personnel
Status: Withdrawn | Type: Observational
Why Stopped: New data published showing EPO to be ineffective in TBI
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Director of Clinical Research, Center for Neuroscience and Regenerative Medicine; Professor of Neurology, Uniformed Services University of the Health Sciences
Other Study IDs: ERMS# 12lO9006; NEU-92-1855 (Other: USUHS)
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Dementia; Traumatic Brain Injury (TBI); Mild Cognitive Impairment (MCI); Chronic Traumatic Encephalopathy (CTE); Post-traumatic Stress Disorder (PTSD)
Keywords: Dementia; Traumatic brain injury (TBI); Mild cognitive impairment (MCI); Chronic traumatic encephalopathy (CTE); Remote effects of TBI; Post-traumatic stress disorder (PTSD_
MeSH Terms: conditions — Dementia; Brain Injuries, Traumatic; Cognitive Dysfunction; Chronic Traumatic Encephalopathy; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- History of TBI: The history of TBI will be assessed by the subject's answers to the Ohio State University Traumatic Brain Injury Identification Method Short Form (OSU TBI-ID SF).
- No history of TBI: The history of TBI will be assessed by the subject's answers to the Ohio State University Traumatic Brain Injury Identification Method Short Form (OSU TBI-ID SF).

SUMMARY:
The objective of this study is to measure the frequency and clinical types of mild cognitive impairment (MCI) or dementia that occur among up to 150 military retirees with and without a history of traumatic brain injury (TBI) among residents of the Armed Forces Retirement Home, Washington D.C. and the Veterans Home of California-Yountville. Investigators will compare the characteristics of dementia in those who have had a prior TBI to the characteristics in those without a history of TBI. It is our hypothesis that the dementia or MCI among those with prior TBI has distinct neuropsychological features that distinguishes it from those with dementia or MCI without a history of TBI.

DETAILED DESCRIPTION:
75 participants with a history of TBI will be the cases (exposed) group. A control group of 75 retirement home residents without a history of TBI who are age-matched to the cases will also be recruited. Participants will be evaluated in a single visit, which will include neurological, psychiatric, and cognitive assessment. The evaluation will take approximately 4 hours. In some cases, the evaluation may be split into two 2 hour sessions.

ELIGIBILITY:
Inclusion Criteria:

Cases (with a history of TBI):

1. Ages 50-95 years
2. History of traumatic brain injury of sufficient severity to have resulted in medical attention (ascertained via the Ohio State University TBI Identification Questionnaire-OSU TBI-ID, and based on DoD/VA criteria)
3. Residence in AFRH-Washington D.C. or the Veterans Home of California-Yountville
4. MMSE score ≥ 20
5. Capacity to provide consent to participate in research (assessment made by study physician)
6. Ability to read and write English

Controls (without a history of TBI):

1. Ages 50-95 years
2. No history of traumatic brain injury of sufficient severity to have resulted in medical attention (ascertained via the Ohio State University TBI Identification Questionnaire-OSU TBI-ID)
3. Residence in AFRH-Washington or the Veterans Home of California-Yountville
4. MMSE score ≥ 20
5. Capacity to provide consent or assent to participate in research
6. Ability to read and write English -

Exclusion Criteria:

Cases (with a history of TBI):

1. History of penetrating brain injury
2. History of disabling neurological or psychiatric condition such as epilepsy (besides posttraumatic epilepsy), multiple sclerosis, cortical stroke, hypoxic-ischemic encephalopathy, encephalitis, or schizophrenia

Controls (without a history of TBI):

History of disabling neurological or psychiatric condition such as epilepsy, multiple sclerosis, cortical stroke, hypoxic-ischemic encephalopathy, encephalitis, or schizophrenia

-

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be recruited from the Armed Forces Retirement Home (AFRH) in Washington, DC and the Veterans Home of California- Yountville. Up to 150 AFRH residents from both the independent living and the assisted living facilities will be invited to take the screening questionnaire and enroll in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dementia or MCI in the two groups (TBI versus no TBI) | Single visit, 4 hours.
  The primary outcome will be the prevalence of dementia/MCI in the two groups (i.e. those with and without a TBI).

SECONDARY OUTCOMES:
Characterization of the types of dementia or MCI that occur in the two groups (TBI or no TBI) | Single visit, 4 hours.
  The characterization of the dementia and cognitive impairment within the two groups based on the neuropsychological testing will be secondary outcomes of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, M.D., Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences; Kristine Yaffe, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - California Veterans Home-Yountville, Yountville, California
  - Armed Forces Retirement Home, Washington D.C., District of Columbia